CLINICAL TRIAL: NCT04784806
Title: Amino Acid Profile and Muscle Protein Synthetic Response to Consuming Meat or Plant-based Alternatives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1548896
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Healthy
Keywords: Meat protein; Plant protein; Muscle protein synthesis
MeSH Terms: interventions — Soy Foods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Consumption of ground beef (Experimental): Consuming 106g of cooked ground beef (85% lean) to deliver 20g of protein.
  Interventions: Other: Ground beef; Other: Ground pork; Other: Tofu; Other: Beyond Meat
- Consumption of ground pork (Experimental): Consuming 118g of cooked ground pork (72% lean) to deliver 20g of protein.
  Interventions: Other: Ground beef; Other: Ground pork; Other: Tofu; Other: Beyond Meat
- Consumption of tofu burger (Experimental): Consuming 113g of cooked tofu to deliver 20g of protein.
  Interventions: Other: Ground beef; Other: Ground pork; Other: Tofu; Other: Beyond Meat
- Consumption of Beyond Meat burger (Experimental): Consuming 113g of Beyond Meat burger to deliver 20g of protein.
  Interventions: Other: Ground beef; Other: Ground pork; Other: Tofu; Other: Beyond Meat

INTERVENTIONS:
Other: Ground beef — Subjects will consume a 106g patty of cooked ground beef.
Other: Ground pork — Subjects will consume a 118g patty of cooked ground pork
Other: Tofu — Subjects will consume a 113g patty of cooked tofu
Other: Beyond Meat — Subjects will consume a 113g BeyondMeat patty.

SUMMARY:
The purpose of the study is to quantify and compare the serum amino acid profile, and muscle protein synthesis rates, in response to consuming isonitrogenous amounts of ground meat (beef and pork) or plant-based alternatives -(soy and pea protein-based patties).

Specific aim 1: Describe the post-prandial amino acid profile in serum in the 3 hours following consumption of the following four burger patties, in quantities calculated to deliver 20 grams of protein: ground beef, ground pork, Beyond Meat® burger, and tofu burger.

Specific aim 2: Compare the ability of these four different foods to activate mTORC1 and protein synthesis in muscle.

DETAILED DESCRIPTION:
Study design:

The first visit will be a brief meeting conducted over Zoom with one of the investigators (Karine Schaal), who will go over the study details with the volunteer, answer their questions, and obtain informed consent. Subjects will sign the informed consent electronically, using DocuSign. Subjects will be given a copy of their signed informed consent form. A paper copy of the consent form will be kept in a locked file cabinet in the office of the principal investigator.

Study volunteers will come to the CTSC Clinical Research Center (CCRC) on four separate occasions. The CCRC is located in the Cypress Building adjacent to the UC Davis Medical Center (2221 Stockton Blvd, Suite D, Sacramento CA 95817).

The four study visits will be test visits scheduled over a two week period (i.e. twice per week for 2 weeks), at the same time in the morning following and overnight (> 12 hour) fast. They will be asked to refrain from vigorous exercise, caffeine, nicotine and alcohol for 24 hours prior to each visit. Female volunteers will be asked to schedule their study visits within the first two weeks of their menstrual cycle (starting on the first day of menstrual bleeding), in order to control for ovarian hormone fluctuations which may impact digestion and metabolism.

Upon arrival to the CCRC on the first test visit, each volunteer's height and weight will be measured.

I. Baseline blood draw. Subjects will then be placed in individual testing rooms, equipped with a reclining phlebotomy armchair. A registered nurse or nurse practitioner will insert a 22G catheter in a forearm vein and an initial 3.5 mL baseline blood sample will be collected.

II. Test meal.

After the baseline blood sample is collected, subjects will consume one of the following four burgers in isonitrogenous amounts to deliver 20 g of protein:

* 106g ground beef patty (85% lean + 15% fat)
* 118g ground pork (72.5% lean + 27.5% fat)
* 113g Beyond Meat® patty
* 113g tofu patty

Each food will be weighed before cooking. The beef, pork and Beyond® burgers will be grilled on an indoor electric grill until internal temperature reaches 165°F to comply with the USDA Recommendations for Food Safety (beef and pork, minimum 160°F) and manufacturer instructions (Beyond Meat®). Tofu burgers are pre-cooked and will be warmed by grilling for 2 minutes, per manufacturer recommendations. The internal temperature of the burgers will be monitored using a meat thermometer. The burgers will be served to the volunteers as soon as they are finished cooking.

Subjects will be asked to consume each patty without buns or condiments within a 10 minute period, and instructed to chew thoroughly. They will also be asked to drink a 6 ounce glass of water with the meal.

III. Postprandial blood draws.

Following consumption of the test meal, the participants will remain at the research site, in their individual testing room, for another 3 hours, sitting quietly - they may bring books or electronic devices to pass the time. Five more blood samples of 3.5 mL each will be obtained at 30, 60, 90, 120 and 180 minutes after the test meal, totaling six blood draws of 3.5mL per visit (21mL per visit), and 84 mL of blood drawn in total for each subject completing the entire study.

Blood will be collected in 3.5 mL serum separating tubes. Approximately 50 microliters of whole-blood will be used to measure blood glucose within 5 minutes of the draw. The rest will be allowed to clot for 1hr before centrifugation at 1000 x g for 10 minutes.The serum will be frozen and kept at -80°C until processed. 100 microliters of each serum sample will be used for determining amino acid concentrations by high performance liquid chromatography (HPLC) at the UC Davis Proteomics Core. Another 100 microliters will be used to measure insulin concentrations via enzyme-linked immunoassay. The rest of the serum will be used for developing the mTORC1 bioassay.

The order in which subjects receive each test meal will be randomized to avoid any order effect, and at least a two-day washout period will be given between visits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy active male (n=8) and female (n=8) volunteers aged 18 - 30 years
* normal weight (BMI between 18 and 25 kg/m2) will be recruited to participate in the study.
* To be considered active, volunteers must meet the following American College of Sports Medicine's guideline for physical activity for healthy adults: performing at least 150 minutes per week of moderate-to-vigorous intensity physical activity.

Exclusion Criteria:

* Health or dietary restriction that would be affected by the foods consumed.
* Known food allergy to legumes (soybeans, peas, peanuts) or meat (beef or pork)
* Anemia (low red blood cell count)
* Overweight or obesity (BMI > 25 kg/m2)
* Currently not meeting the ACSM physical activity recommendations (IPAQ score < 150 min/week of moderate-to-vigorous physical activity)
* Metabolic or endocrine disorder that would affect the digestion, absorption, and/or physiological response to any of the nutrients ingested
* Receiving any medication that may interfere with the study
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Quantification of serum amino acid concentrations after consuming each test meal. | Baseline and 30, 60, 90, 120 and 180 minutes after consuming each test meal
  A fasted 3.5mL baseline blood sample will be collected in serum separating tubes, after which subjects will consume one of the four patties. Five 3.5mL blood samples will be obtained at 30, 60, 90, 120 and 180 minutes following the patty consumption.
  Blood will be allowed to clot for 1hr before centrifugation at 1000 x g for 10 minutes. The serum will be frozen and kept at -80°C until processed. 100 microliters of each serum sample will be used for determining amino acid concentrations by high performance liquid chromatography (HPLC) at the UC Davis Proteomics Core.
Quantification of muscle protein synthesis rates in vitro | Baseline and 30, 60, 90, 120 and 180 minutes after consuming each test meal
  The rest of the serum obtained from the procedures described in Outcome 1 will be used for developing the mTORC1 bioassay and quantify the rate of muscle protein synthesis in vitro.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Baar, Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- CTSC Clinical Research Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang JE, Moore DR, Kujbida GW, Tarnopolsky MA, Phillips SM. Ingestion of whey hydrolysate, casein, or soy protein isolate: effects on mixed muscle protein synthesis at rest and following resistance exercise in young men. J Appl Physiol (1985). 2009 Sep;107(3):987-92. doi: 10.1152/japplphysiol.00076.2009. Epub 2009 Jul 9. PMID 19589961
- [Background] Dickinson JM, Fry CS, Drummond MJ, Gundermann DM, Walker DK, Glynn EL, Timmerman KL, Dhanani S, Volpi E, Rasmussen BB. Mammalian target of rapamycin complex 1 activation is required for the stimulation of human skeletal muscle protein synthesis by essential amino acids. J Nutr. 2011 May;141(5):856-62. doi: 10.3945/jn.111.139485. Epub 2011 Mar 23. PMID 21430254
- [Background] Baar K, Esser K. Phosphorylation of p70(S6k) correlates with increased skeletal muscle mass following resistance exercise. Am J Physiol. 1999 Jan;276(1):C120-7. doi: 10.1152/ajpcell.1999.276.1.C120. PMID 9886927
- [Background] Witard OC, McGlory C, Hamilton DL, Phillips SM. Growing older with health and vitality: a nexus of physical activity, exercise and nutrition. Biogerontology. 2016 Jun;17(3):529-46. doi: 10.1007/s10522-016-9637-9. Epub 2016 Feb 15. PMID 26878863
- [Background] Wolfson RL, Sabatini DM. The Dawn of the Age of Amino Acid Sensors for the mTORC1 Pathway. Cell Metab. 2017 Aug 1;26(2):301-309. doi: 10.1016/j.cmet.2017.07.001. PMID 28768171
- [Background] van Vliet S, Burd NA, van Loon LJ. The Skeletal Muscle Anabolic Response to Plant- versus Animal-Based Protein Consumption. J Nutr. 2015 Sep;145(9):1981-91. doi: 10.3945/jn.114.204305. Epub 2015 Jul 29. PMID 26224750
- [Background] Tipton KD, Ferrando AA, Phillips SM, Doyle D Jr, Wolfe RR. Postexercise net protein synthesis in human muscle from orally administered amino acids. Am J Physiol. 1999 Apr;276(4):E628-34. doi: 10.1152/ajpendo.1999.276.4.E628. PMID 10198297
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-the-effect-of-meat-or-plant-based-alternatives-on-muscles-574019/